CLINICAL TRIAL: NCT02432170
Title: Weight-Bearing Tomosynthesis In Evaluation of Foot/AnkIe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Alice Ha, Associate Professor, Radiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 48992
Record Dates: First submitted 2015-04-15; First posted 2015-05-04 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foot/Ankles imaged with tomosynthesis (Experimental): Intervention: Digital Tomosynthesis of Foot and Ankle
  The intervention, digital tomosynthesis of the foot and ankle, will be done on eligible participants. The resulting images will be compared to radiography and weight-bearing CT images from the same participants.
  Interventions: Device: Digital Tomosynthesis of Foot and Ankle

INTERVENTIONS:
Device: Digital Tomosynthesis of Foot and Ankle — Imaging Technique

SUMMARY:
This study aims to compare digital tomosynthesis with radiography and weight-bearing CT as an imaging technique to assess arthritis in the foot and ankle.

DETAILED DESCRIPTION:
The overall goal of this study is to improve radiologic evaluation of foot and ankle arthritis. Today's standard of care, radiography, provides limited two-dimensional evaluation of joint alignment, arthritic changes, posttraumatic changes, and congenital deformities due to overlapping bone densities. Evaluation is even more limited in post-surgical patients due to overlapping metallic hardware. Computed tomography (CT), the current problem-solving tool, offers more "level-by-level" three dimensional information, but is fraught with additional cost, additional radiation dose, beam-hardening artifacts from hardware, and the need for additional equipment. Most importantly, patients are not weight-bearing during conventional CT, therefore masking the true extent of malalignment or arthritic joint space narrowing. At the University of Washington, physicians attempt to overcome the last problem by performing simulated weight-bearing CT. The study proposes an alternate solution to this problem using a novel application of an old method, digital tomosynthesis. Specific aims of the study are 1) to compare radiography, tomosynthesis, and simulated-weight bearing CT in their ability to detect foot/ankle malalignment, 2) to compare the abilities of these three modalities to detect arthritis changes such as joint space narrowing, osteophytes, and subchondral cysts, and 3) to compare their abilities to detect bony deformities such as acute fracture, old fracture deformity, or partial fusion (post traumatic or post surgical). Radiographic assessment will be correlated with clinical outcome using clinical notes and functional outcome such as the Lower Extremity Functional Scale (LEFS) questionnaire. Successful results from this initial study will have the potential to change practice paradigm in how to image foot and ankle arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. adult age (18 years or older)
2. clinical orthopedic surgery follow-up notes available at University of Washington
3. ability to complete the Lower Extremity Functional Scale (LEFS) or equivalent questionnaire at the time of the study, a well established survey to test for functional ability in lower extremity

Exclusion Criteria:

1. inability to use the simulated weight bearing CT machine due to pain
2. prior complete osseous fusion of foot/ankle joints
3. prior total ankle arthroplasty
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Severity of Arthritis (assessed through reading radiologic images and through a pain survey) | One day
  Severity of arthritis will be assessed through reading radiologic images and through a pain survey filled out by participants.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States